CLINICAL TRIAL: NCT02330627
Title: Positive Valence System Enhancement Treatment for Anxiety and Depression: Clinical Efficacy and Neural Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Charles Taylor, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5UL1TR000100 (NIH); 5UL1TR000100 (NIH)
Record Dates: First submitted 2014-12-24; First posted 2015-01-05 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Anxiety Disorders and Symptoms; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive Valence System Treatment (Experimental): 10 one-hour individual sessions comprised of psychoeducation and positive activity interventions designed to increase positive emotions, cognitions, and behaviors.
  Interventions: Behavioral: Positive Valence System Treatment
- Delayed Treatment (Waitlist) (No Intervention)

INTERVENTIONS:
Behavioral: Positive Valence System Treatment — Clinician-administered one-hour treatment sessions focused on presenting rationale and instructions for completing positive activity exercises (e.g., gratitude, acts of kindness) between sessions.
  Arms: Positive Valence System Treatment

SUMMARY:
The proposed project aims to test the efficacy and neural correlates of a behavioral treatment program comprised of positive activity interventions in a sample of individuals seeking treatment for anxiety or depression. Participants will be randomly assigned to an immediate or delayed treatment condition, and will be compared on measures of positive and negative emotions, brain responses to reward and punishment/loss, subjective well-being, and symptoms at baseline and post-treatment.

DETAILED DESCRIPTION:
Current treatment approaches for anxiety and depression emphasize the reduction of negative emotions and distress as the central goal of treatment. However, these conditions are also characterized by low levels of positive emotions, which, although fundamental for life satisfaction and well-being, have traditionally not been a focus of treatment. The proposed project aims to test the efficacy of an integrated treatment regimen designed to modulate functioning of core component processes of the positive emotion system. Specifically, we will implement positive emotion enhancement procedures, previously tested and validated in non-clinical samples (Huffman et al., 2011; Lyubomirsky et al., 2005), in a broad community sample of n=30 individuals seeking treatment for anxiety or depression. Participants will be randomly assigned to a multi-session positive valence system targeted treatment (n=15) or a waitlist control group (n=15). Participants will be assessed at baseline and post-treatment and compared on measures of positive and negative emotions, brain responses to reward and punishment/loss, subjective well-being, and symptoms. Aim 1 will test the hypothesis that participants assigned to the positive emotion enhancement intervention will display greater increases in positive affect and enhanced activity in neural systems that regulate responses to reward (e.g., nucleus accumbens) relative to participants in the waitlist control group. Aim 2 will explore whether the effects of the positive emotion system treatment generalize to parallel measures of the negative emotion system (i.e., negative affect and neural reactivity to aversive outcomes). We will also explore the effects of the intervention on subjective well-being and life satisfaction, and will examine the relationship between changes in subjective emotions and neural indices of positive and negative valence functioning with changes in well-being and life satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Score on the PHQ-9 is 10 or higher and/or score on the OASIS is 8 or higher.
2. Between the ages of 18-55, inclusive.
3. Have sufficient proficiency in the English language to understand and complete interviews, questionnaires, and all other study procedures.

Exclusion Criteria:

1. No telephone or easy access to telephone.
2. Any substance use disorder in the past year except subjects with mild alcohol, nicotine, caffeine, and marijuana use disorders will be permitted in the study.
3. Bipolar I or Psychotic disorders.
4. Moderate to severe traumatic brain injury with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study.
5. Current and regular use (more days than not during the past 30 days) of a medication that could affect brain functioning, such as anxiolytics, antipsychotics, antidepressants, mood stabilizers, beta-blockers, sleep medications, opioids/codeine, migraine medications.
6. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60 minutes; prior neurosurgery; tattoos with metal dyes, unwillingness to remove body piercings, and pregnancy.
7. non-correctable vision or hearing problems, as some tests require intact sensory functioning.
8. Concurrent psychosocial treatment: Participants completing ongoing psychosocial treatment will be required to meet a 12-week stability criteria so that symptom changes as a result of other psychosocial treatments are not confounded with changes due to the research.
9. Inability to complete the initial assessment battery or treatment sessions.
10. Clinical conditions assessed by the interviewer that necessitate more imminent clinical care (e.g., active suicidal ideation). These criteria are in place so participants with these other, more several symptoms can be referred for appropriate mental health services.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles T Taylor, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Psychiatry Clinical Research, La Jolla, California, United States

REFERENCES:
- [Result] Taylor CT, Lyubomirsky S, Stein MB. Upregulating the positive affect system in anxiety and depression: Outcomes of a positive activity intervention. Depress Anxiety. 2017 Mar;34(3):267-280. doi: 10.1002/da.22593. Epub 2017 Jan 6. PMID 28060463
- [Derived] Kryza-Lacombe M, Spaulding I, Ku CK, Pearson N, Stein MB, Taylor CT. Amplification of positivity for depression and anxiety: Neural prediction of treatment response. Behav Res Ther. 2024 Jul;178:104545. doi: 10.1016/j.brat.2024.104545. Epub 2024 Apr 23. PMID 38714105
- [Derived] Kryza-Lacombe M, Pearson N, Lyubomirsky S, Stein MB, Wiggins JL, Taylor CT. Changes in neural reward processing following Amplification of Positivity treatment for depression and anxiety: Preliminary findings from a randomized waitlist controlled trial. Behav Res Ther. 2021 Jul;142:103860. doi: 10.1016/j.brat.2021.103860. Epub 2021 Apr 15. PMID 33894554
- [Derived] Taylor CT, Pearlstein SL, Kakaria S, Lyubomirsky S, Stein MB. Enhancing Social Connectedness in Anxiety and Depression Through Amplification of Positivity: Preliminary Treatment Outcomes and Process of Change. Cognit Ther Res. 2020 Aug;44(4):788-800. doi: 10.1007/s10608-020-10102-7. Epub 2020 Apr 19. PMID 32661447
- See also: Upregulating the positive affect system in anxiety and depression: Outcomes of a positive activity intervention. — http://www.ncbi.nlm.nih.gov/pubmed/28060463

RESULTS

PARTICIPANT FLOW:
Groups:
- Delayed Treatment (Waitlist): No treatment received for 10 weeks
Period: Overall Study
Arm/Group | Positive Valence System Treatment | Delayed Treatment (Waitlist)
Started | 16 | 13
Completed | 15 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the delayed treatment (waitlist) arm initiated an alternate treatment following the pre-assessment and was thus excluded from the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Valence System Treatment | Delayed Treatment (Waitlist) | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (12.2) | 29.0 (12.0) | 29.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 13 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 12 | 8 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive Affect (Positive and Negative Affect Schedule; Modified Differential Emotions Scale; Composite)
Description: The Positive and Negative Affect Schedule (PANAS) measures positive affect. Items are answered on a 5 point scale, 1 (Very slightly or not at all) to 5 (Extremely). The positive affect scale ranges from 10-50 and higher scores indicate greater levels of positive affect.
  The Modified Differential Emotions Scale (mDES) measures positive emotions. Items are answered on a 5 point scale, 0 (Never/Not at all) to 4 (Most of the time/Extremely). Higher scores on the positive emotions sub-scale indicate higher levels of positive emotion.
  Participants' scores on the PANAS and mDES were first standardized across assessment sessions by converting to Z scores (M=0, SD=1) across both groups. The composite index of positive affect at each assessment point was the mean of the Z scores for that occasion. Higher z-scores indicate an increase in positive affect from baseline to post-treatment.
Time Frame: Baseline, 10 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Positive Valence System Treatment | Delayed Treatment (Waitlist)
Number analyzed (Participants) | 16 | 12
z-score
  Pre-assessment | -0.41 (.96) | -0.40 (.54)
  Post-assessment | 0.73 (.87) | -0.02 (.79)

2. Primary Outcome: Change From Baseline in Blood Oxygen Level Dependent (BOLD) Response in the Striatum and Medial Prefrontal Cortex, as Measured With Functional Magnetic Resonance Imaging (fMRI) During Reward Trials on the Monetary Incentive Delay (MID) Task
Description: Change from pre- to post-assessment in neural activation during reward trials on the MID task.
Time Frame: Baseline, 10 weeks
Reporting Status: Not Posted, anticipated posting 2022-03

3. Secondary Outcome: Change From Baseline in Negative Affect (Positive and Negative Affect Schedule; Modified Differential Emotions Scale; Composite)
Description: The Positive and Negative Affect Schedule (PANAS) measures negative affect. Items are answered on a 5 point scale, 1 (Very slightly or not at all) to 5 (Extremely). The negative affect scale ranges from 10-50 and lower scores indicate lower levels of negative affect.
  The Modified Differential Emotions Scale (mDES) measures negative emotions. Items are answered on a 5 point scale, 0 (Never/Not at all) to 4 (Most of the time/Extremely). Lower scores on the negative emotions sub-scale indicate lower levels of negative emotion.
  Participants' composite scores on the PANAS and mDES were first standardized across assessment sessions by converting to Z scores (M=0, SD=1) across both groups. The composite index of negative affect at each assessment point (i.e., pre assessment - at baseline, post assessment - 10 weeks after baseline) was the mean of the Z scores for that occasion. Lower z-scores indicate a decrease in negative affect from baseline to post-treatment.
Time Frame: Baseline, 10 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Positive Valence System Treatment | Delayed Treatment (Waitlist)
Number analyzed (Participants) | 16 | 12
z-score
  Pre Assessment | 0.17 (0.62) | 0.70 (0.89)
  Post Assessment | -0.19 (0.40) | 0.29 (1.11)

4. Secondary Outcome: Change From Baseline in Blood Oxygen Level Dependent (BOLD) Response in the Striatum and Insula, as Measured With Functional Magnetic Resonance Imaging (fMRI) During Loss Trials on the Monetary Incentive Delay (MID) Task
Description: Change from pre- to post-assessment in neural activation during loss trials on the MID
Time Frame: Baseline, 10 weeks
Reporting Status: Not Posted, anticipated posting 2022-03

5. Other Pre Specified Outcome: Change From Baseline in Quality of Life and Well-being (Composite of Quality of Life, Enjoyment, and Satisfaction Questionnaire; Satisfaction With Life Scale)
Description: The Quality of Life, Enjoyment, and Satisfaction Questionnaire (Q-LES-Q) measures the degree of satisfaction experienced by participants in various areas of daily functioning. Items are rated on a 5 point scale, 1 (Very Poor) to 5 (Very Good). The scale ranges from 14-70; higher scores indicate higher levels of life satisfaction.
  The Satisfaction With Life Scale (SWLS) measures global cognitive judgments of one's life satisfaction. Items are rated on a 7 point scale, 1 (Strongly Disagree) to 7 (Strongly Agree). The scale ranges from 5-35; higher scores indicate higher levels of life satisfaction.
  Participants' scores on the Q-LES-Q and the SWLS were first standardized across assessment sessions by converting to Z scores (M=0, SD=1) across both groups. The composite index of quality of life and well-being at each assessment point was the mean of the Z scores for that occasion. Higher z-scores indicate an increase in quality of life and well-being from baseline to post-treatment.
Time Frame: Baseline, 10 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Positive Valence System Treatment | Delayed Treatment (Waitlist)
Number analyzed (Participants) | 16 | 12
z-score
  Pre-assessment | -.25 (.77) | -.34 (.81)
  Post-assessment | .76 (.81) | -.35 (.87)

6. Other Pre Specified Outcome: Change From Baseline in Anxiety (Overall Anxiety Severity and Impairment Scale; State Trait Anxiety Inventory - Trait Composite)
Description: The Overall Anxiety Severity and Impairment Scale (OASIS) measures frequency, severity, and functional impairment of anxiety symptoms. Items are rated on a 4 point scale, 0 (None) to 4 (Extreme). The scale ranges from 0-20 and higher scores indicate higher levels of anxiety.
  The State Trait Anxiety Inventory - Trait (STAI-T) measures general anxiety. Items are rated on a 4 point scale, 1 (Almost Never) to 4 (Almost Always). The scale ranges from 20-80 and higher scores indicate higher levels of anxiety.
  Participants' composite scores on the OASIS and the STAI were first standardized across assessment sessions by converting to Z scores (M=0, SD=1) across both groups. The composite index of anxiety at each assessment point (i.e., pre assessment - at baseline, post assessment - 10 weeks after baseline) was the mean of the Z scores for that occasion. Lower z-scores indicate a decrease in anxiety from baseline to post-treatment.
Time Frame: Baseline, 10 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Positive Valence System Treatment | Delayed Treatment (Waitlist)
Number analyzed (Participants) | 16 | 12
z-score
  Pre Assessment | .14 (.54) | .40 (.62)
  Post Assessment | -.61 (.68) | .23 (.91)

7. Other Pre Specified Outcome: Change From Baseline in Depression (Patient Health Questionnaire-9; Beck Depression Inventory-II Composite)
Description: The Patient Health Questionnaire-9 (PHQ-9) measures depression symptoms. Items are rated on a 4 point scale, 0 (Not at all) to 3 (Nearly every day). The scale ranges from 0-27 and higher scores indicate higher levels of depression.
  The Beck Depression Inventory-II (BDI-II) measures the severity of depression. Participants choose 1 of 4 response options; a value of 0 to 3 is assigned to each response option. The scale ranges from 0-63 and higher scores indicate higher severity of depression.
  Participants' composite scores on the PHQ-9 and the BDI-II were first standardized across assessment sessions by converting to Z scores (M=0, SD=1) across both groups. The composite index of depression at each assessment point (i.e., pre assessment - at baseline, post assessment - 10 weeks after baseline) was the mean of the Z scores for that occasion. Lower z-scores indicate a decrease in depression from baseline to post-treatment.
Time Frame: Baseline, 10 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Positive Valence System Treatment | Delayed Treatment (Waitlist)
Number analyzed (Participants) | 16 | 12
z-score
  Pre Assessment | .29 (.90) | .47 (.77)
  Post Assessment | -.87 (.55) | .29 (.97)

ADVERSE EVENTS:
Arm/Group | Positive Valence System Treatment | Delayed Treatment (Waitlist)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 0/16 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No